CLINICAL TRIAL: NCT04823624
Title: TIM3 Inhibition With MBG453 for Patients With Lower Risk MDS: an Adaptive Two-Stage Phase II Clinical Trial
Brief Title: MBG453 in Lower Risk MDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Andrew Mark Brunner, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-637
Record Dates: First submitted 2021-03-09; First posted 2021-04-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — sabatolimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MG MBG453 (Experimental): Participants will be given MBG453 On Day 1 of each cycle 28 days (4 weeks) study cycle
  Interventions: Drug: MBG453

INTERVENTIONS:
Drug: MBG453 — intravenous infusion

SUMMARY:
This research study is assessing the efficacy of MBG-453, a humanized monoclonal antibody, in treating myelodysplastic syndromes (MDS).

The name of the study drug involved in this study is MBG453.

DETAILED DESCRIPTION:
This is an adaptive two-stage phase II clinical trial to assess the activity of the anti-TIM-3, (T cell immunoglobulin domain and mucin domain) antibody, MBG453, in patients with lower-risk myelodysplastic syndromes (MDS), not eligible for or progressing on frontline therapy.

The U.S. Food and Drug Administration (FDA) has not approved MBG453 for myelodysplastic syndromes (MDS), but it has been approved for other uses.

The study drug (MBG453) may interact with TIM-3 (an antibody which is a protein that attaches to foreign infectious/invading cells and signals the immune system) which might aid the immune system's response by helping immune cells recognize, find, and destroy cancer cells in the body.

The research study procedures include screening for eligibility and study treatment, including evaluations and follow up visits.

Participants will receive study treatment for as long as they and their doctor believe they are benefiting from the study drug. Participants will then be followed for 12 months after their last dose of the study drug or until they withdraw their consent to be contacted.

It is expected that about 20 people will take part in this research study

ELIGIBILITY:
Inclusion Criteria:

* Lower risk MDS patients (IPSS-R score ≤ 3.5 at diagnosis) who have progressed or are refractory to/intolerant of prior therapy and meet one of the following categories:

  * RBC transfusion dependent according to IWG criteria must either be unresponsive to prior ESA therapy or have an EPO level > 500
  * Prior HMA therapy
  * Patients with the following cytopenias who otherwise are felt to require treatment per the treating physician:

    * Platelets < 50k/uL
    * ANC < 500 cells/uL
  * Patients with MDS with isolated del(5q) ("5q- syndrome") must have progressed on or not tolerated lenalidomide
  * Patients who are not felt to be candidates for or lack other standard treatment options. Patients with prior luspatercept exposure are eligible.
  * Patients with dysplastic type CMML (WBC < 13,000 cells/uL) meeting the above criteria are eligible; responses will be assessed using MDS criteria
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of MGB453 in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG performance status ≤2 (see Appendix A).
* Participants must have adequate organ and marrow function as defined below within 21 days of treatment:

  * Total bilirubin ≤ 2 mg/dL (unless due to Gilbert's in which case it must be <3 mg/dL)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * Creatinine clearance ≥30 mL/min/1.73 m2 (by MDRD calculation)
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load over the prior 6 months are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had chemotherapy or radiotherapy within 14 days or five half-lives, whichever is shorter, prior to the first dose of study treatment.
* Participants who are receiving any other investigational agents; a washout of 14 days or 5 half-lives, whichever is longer, is required. The washout period for biologic agents should be 28 days since the last dose.
* Prior exposure to a TIM-3 inhibitor.
* Active autoimmune disease requiring > 10 mg per day of prednisone or the equivalent. Inactive or controlled autoimmune disease is allowed.
* Prior solid organ transplant is exclusionary. Patients with prior hematopoietic cell transplant are eligible if they are over 6 months from transplant and not on any related immunosuppressive therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MBG453.
* Active untreated or concurrent malignancy that is distinct in primary site or histology, excluding:

  * The following will not be exclusionary: non-melanoma skin cancer, noninvasive colonic polyps, superficial bladder tumors, cervical cancer in-situ, ductal carcinoma in situ of the breast, monoclonal B-cell lymphocytosis, or monoclonal gammopathy of undetermined significance.
  * Hormonal therapy is allowed.
  * History of other malignancy is allowed if not requiring active management.
  * Other malignancies that were treated with curative intent at least 1 year prior to study screening and without evidence of active disease will be allowed.
  * Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial pending discussion with the principal investigator.
* Participants with uncontrolled intercurrent illness.
* Participants must not have clinically active HBV or HCV; testing is not required
* Receipt of a live vaccination within 28 days of cycle 1 day 1
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Female contraception is required. Pregnant women are excluded from this study because MBG453 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MBG453, breastfeeding should be discontinued. Women of child-bearing potential should use highly effective methods of contraception during treatment and for 150 days after the last dose of MBG453.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 6 months
  Assessed on the proposal for the modification of the International Working Group (IWG) response criteria in myelodysplasia (Cheson et al., 2006), but modified to include complete remission with partial hematologic improvement CRh (Bloomfield et al., 2018), and the 2018 proposed update for hematologic responses and transfusion independence (TI) (Platzbecker et al., 2019). Patients with dysplastic-type CMML will use MDS risk-stratification and response assessment criteria.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | during the intervention, an average of 1 year
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade.
Overall survival (OS) 1-year | 1 year
  Estimated using the Kaplan and Meier method.
Progression free survival (PFS) | through study completion, an average of 1 year
  Estimated using the Kaplan and Meier method.
Time to disease progression | through study completion, an average of 1 year
  Estimated using the Kaplan and Meier method.
Duration of response | through study completion, an average of 1 year
  Estimated using the Kaplan and Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Brunner, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT04823624/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT04823624/ICF_001.pdf